CLINICAL TRIAL: NCT05125120
Title: THE EFFECT OF THE COGNITIVE ORIENTATION TO DAILY OCCUPATIONAL PERFORMANCE (CO-OP) APPROACH IN CHILDREN WITH ATTENTION DEFICIT AND HYPERACTIVITY DISORDER ON MOTOR PERFORMANCE AND EXECUTIVE FUNCTIONS: A RANDOMIZED CONTROLLED STUDY
Brief Title: THE EFFECT OF THE COGNITIVE ORIENTATION TO DAILY OCCUPATIONAL PERFORMANCE (CO-OP) APPROACH IN CHILDREN WITH ATTENTION DEFICIT AND HYPERACTIVITY DISORDER ON MOTOR PERFORMANCE AND EXECUTIVE FUNCTIONS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SEDANUR GÜRLEK, SEDANUR GÜRLEK (Master's degree)(Occupational Therapist), Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HU.SGURLEK.001
Record Dates: First submitted 2021-10-24; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Cognitive Orientation; Executive Dysfunction; Motor Activity
MeSH Terms: conditions — Orientation, Spatial; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Attention Deficit and Hyperactivity Disorder (Other): Attention Deficit and Hyperactivity Disorder (CO-OP Group) Attention Deficit and Hyperactivity Disorder (Control Group)
  Interventions: Other: COGNİTİVE ORİENTATİTON DAİLY OCCUPATİONAL PERFORMANCE APPROACH

INTERVENTIONS:
Other: COGNİTİVE ORİENTATİTON DAİLY OCCUPATİONAL PERFORMANCE APPROACH — Polatajko et al. (2001) developed the CO-OP approach, which is an occupation-oriented problem-solving approach that combines cognitive strategies to help children acquire motor abilities throughout daily tasks (9, 29). The CO-OP approach of therapy focuses on the goal or task at hand rather than the acquisition of functions in occupational performance. CO-OP is a 'deductive' or 'occupational performance-oriented' approach that focuses on the activity target selected throughout the therapy, as opposed to 'inductive' or 'impairment-focused' alternatives (13). As a verbal approach, CO-OP focuses on skill acquisition at the activity level and strives to provide children with global problem-solving skills. Necessary performance strategies specific to the child and the activity are determined with a customised programme (12, 30). Skill acquisition, cognitive strategy development, and adapting and transferring these acquired skills to daily life are the three key goals of the approach.

SUMMARY:
Attention deficit and hyperactivity disorder (ADHD) is a behavioural and neurodevelopmental disorder that can affect behavioural, emotional, academic, social, and cognitive functions and is not age-appropriate. The prevalence of ADHD among school children is reported to be 3%-11%. Children with ADHD have difficulties paying attention to details, concentrating, completing tasks and following instructions, among other social and academic challenges. In children with ADHD, insufficient activity in the prefrontal regions of the brain has been evidenced, which is linked to executive function skills. Such children have difficulties in performing executive functions that require a high level of cognitive skills, such as self-control and regulation, as well as sequencing and planning tasks. The Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) addresses executive dysfunction as a characteristic of ADHD. At the same time, 45%-70% of these children show problems in motor skills. Motor problems associated with ADHD, such as manual dexterity, bilateral coordination, and postural balance, can lead to difficulty in everyday living tasks, such as eating and writing, as well as social adaptability, academic skills, and peer interactions. For this reason, motor skill problems along with symptoms of inattention, hyperactivity, and impulsivity, should be addressed as part of the treatment strategy. ADHD has an impact on a child's independence for daily activities. As a result, child-specific occupational therapy approaches are critical for the sensory, motor, and cognitive areas that affect children's occupational performance in basic and instrumental activities of daily living, participation, rest and sleep, play, and leisure.

DETAILED DESCRIPTION:
Afyonkarahisar University of Health Sciences Non-Invasive Clinical Research Ethics Committee evaluated the study with the 2011-KAEK-2 ethics committee code. The study was planned to be carried out in Afyonkarahisar State Hospital Occupational Therapy Unit. It was planned to include 30 children between the ages of 7 and 12 who were diagnosed with ADHD according to the DSM-5 criteria by a child psychiatrist. Children will be randomly divided into two groups: 15 in the intervention group and 15 in the control group. At the beginning of the study, the purpose of the study will be explained to the family and the child and informed consent forms will be signed. Standard tests will be applied after the sociodemographic information of the child and his family is obtained. With the CO-OP approach, the intervention group will receive two sessions of therapy per week, each for approximately one hour, for a total of 6 weeks and 12 sessions. After 6 weeks, standard assessments will be repeated. The control group will receive the same standardized assessments at baseline and 6 weeks later with no further intervention.

ELIGIBILITY:
Inclusion criteria:

* The child is between 7 and 12 years old
* Meeting the diagnostic criteria for ADHD
* Continuing drug therapy with methylphenidate
* Attending school

Exclusion Criteria:

* Having a mental, chronic neurological or orthopedic disorder in addition to ADHD

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The Canadian Occupational Performance Measure (COPM) | five weeks
  It is an client-centred semi-structured interview method in which individuals score their performance and satisfaction in the activities that they need, want, or are required to accomplish in the areas of self-care, productivity, and leisure (17, 18). On a 10-point scale (1=not able to do=not satisfied at all, 10=can be done=pleased), the individual ranks the activities that he or she considers significant for themselves separately in terms of performance and satisfaction
Goal Attainment Scaling (GAS) | five weeks
  It is used to determine whether children have met their functional activity goals. It's critical that the objectives are clear, measurable, and well-timed (21, 22). The various achievable results for each aim are defined independently at five levels while scoring the GAS: -2, -1, 0, +1, and +2. The initial level is -2, and the child's level is re-evaluated after the application
The Bruininks-Oseretsky Test of Motor Proficiency and Performance-Short Form (BOTMP-SF) | five weeks
  The BOTMP-SF which was modified from the long version and is used to assess children's motor abilities, has 14 items and a maximum score of 98. BOTMP-SF assesses upper extremity coordination, balance, visual-motor control, and other skills in three areas: gross motor, gross-fine motor, and fine motor
The Executive Functions and Occupational Routines Scale (EFORTS) | five weeks
  This scale is used to assess executive function skills and activity routines of children aged 6-12 years, including impulsivity, verbal and nonverbal memory, self-regulation, planning, and problem-solving. It is divided into three sections: morning-evening routine, game-entertainment routines, and social routines
Visual Analogue Scale (VAS) | five weeks
  The VAS is a scale for converting some values that are difficult to measure numerically into numerical data. The participant uses a vertical line on a 0-10 cm scale to denote his or her emotional state, and the distance is measured with a ruler. The VAS was used to measure the level of satisfaction of families with therapy in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar State Hospital, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Derived] Gurlek S, Bumin G. The effect of cognitive orientation to daily occupational performance in children with attention deficit hyperactivity disorder: A pilot randomized controlled study. Appl Neuropsychol Child. 2024 Jul 31:1-10. doi: 10.1080/21622965.2024.2385679. Online ahead of print. PMID 39081141